CLINICAL TRIAL: NCT02345954
Title: Laparoscopic Supracervical Hysterectomy and Sacropexy Compared to Uterus Conserving Hysteropexy: a Randomized Clinical Trial
Brief Title: Laparoscopic Supracervical Hysterectomy and Sacropexy Versus Hysteropexy Study
Acronym: HysPex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dimitri Sarlos, Chair Department of Gynecology, Kantonsspital Aarau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lapSKPvslapHP
Record Dates: First submitted 2014-11-21; First posted 2015-01-26 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Uterus Prolapse
Keywords: Uterus Prolapse; Laparoscopic Sacropexy; Laparoscopic Hysteropexy
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supracervical Hysterectomy and Sacropexy (Experimental): Laparoscopic Supracervical Hysterectomy and Sacropexy
  Interventions: Procedure: Laparoscopic Supracervical Hysterectomy and Sacropexy
- Hysteropexy (Experimental): Laparoscopic Hysteropexy
  Interventions: Procedure: Laparoscopic Hysteropexy

INTERVENTIONS:
Procedure: Laparoscopic Supracervical Hysterectomy and Sacropexy — Laparoscopic supracervical hysterectomy and laparoscopic sacrocolpopexy
  Arms: Supracervical Hysterectomy and Sacropexy
Procedure: Laparoscopic Hysteropexy — Laparoscopic hysteropexy
  Arms: Hysteropexy

SUMMARY:
The purpose of this study is to compare the operative, anatomic functional outcome as well as the subjective outcome of laparoscopic supracervical hysterectomy and sacropexy compared to laparoscopic hysteropexy (conserving the uterus).

The investigators expect that both laparoscopic procedures are equal in regards to operation time, complication rate, anatomic and functional outcome as well as subjective outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Symptomatic uterus prolapse (uterus < 300g)
* Patient able to sign the informed consent and to fulfil the follow up visits

Exclusion Criteria:

* Indication: Pathologies of the uterus (postmen. bleeding, high endometrium at ultrasound (>5 mm), abnormal PAP smear in the last 5 years, bleeding anomalies in premenopausal patients
* General medical contraindications to a surgical operation

  * tumor/ malignant disease
  * bacterial infection at time of surgery
  * drug or medication abuse at time or just before surfer
* Disease which would make a correct assessment of the patient impossible (e.g. psychiatric condition)
* Known hypersensitivity to the implanted materials
* Immaturity, inability to answer/understand questions
* Planned pregnancy
* Participation to other studies (drugs or medical techniques) which could influence the results of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Operation time | expected average of 150 minutes
  Comparison of operation time in the 2 arms of the study

SECONDARY OUTCOMES:
Intra- and postoperative complication rate | 1 year
Duration of anaesthesia | expected average of 200 minutes
IUGA Pelvic Organ Prolapse Quantification (POP-Q) | 8 weeks before surgical intervention and at follow up 6 weeks, 6 months and 12 months after intervention
Bladder and bowel function, Prolapse symptoms, Sexuality | 8 weeks before surgical intervention and at follow up 6 weeks, 6 months and 12 months after intervention
  Assessed via Pelvic Function Questionnaire
Quality of Life | 8 weeks before surgical intervention and at follow up 6 weeks, 6 months and 12 months after intervention
  EQ-5D-5L questionnaire
Patient satisfaction after surgery | At follow up 6 weeks, 6 months and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, MD, Study Chair — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Aargau (AG), Switzerland

REFERENCES:
- [Background] Sarlos D, Kots L, Stevanovic N, von Felten S, Schar G. Robotic compared with conventional laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2012 Sep;120(3):604-11. doi: 10.1097/AOG.0b013e318265b61a. PMID 22914470
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Khunda A, Vashisht A, Cutner A. New procedures for uterine prolapse. Best Pract Res Clin Obstet Gynaecol. 2013 Jun;27(3):363-79. doi: 10.1016/j.bpobgyn.2012.12.004. Epub 2013 Jan 5. PMID 23298608
- [Background] Krause HG, Goh JT, Sloane K, Higgs P, Carey MP. Laparoscopic sacral suture hysteropexy for uterine prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jun;17(4):378-81. doi: 10.1007/s00192-005-0019-0. Epub 2005 Nov 30. PMID 16319998
- [Background] Price N, Slack A, Jackson SR. Laparoscopic hysteropexy: the initial results of a uterine suspension procedure for uterovaginal prolapse. BJOG. 2010 Jan;117(1):62-8. doi: 10.1111/j.1471-0528.2009.02396.x. PMID 20002370